CLINICAL TRIAL: NCT01124448
Title: Oral Administration of a Probiotic to Lactating Women: Microbiological, Immunological, Transcriptomics and Metabolomics Effects
Brief Title: Global Effects of a Probiotic Strain on Lactating Women
Acronym: PROBIOLAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: National Research Council, Spain (Other Government); University of Valencia (Other); Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Juan M. Rodríguez, Professor, PhD, Universidad Complutense de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PROBIOLAC
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Mastitis
MeSH Terms: conditions — Mastitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus salivarius PS2 (Experimental): Women with mastitis (n=25) receiving Lactobacillus salivarius PS2 (9.5 log per day, 21 days)
  Interventions: Biological: Lactobacillus salivarius PS2
- Lactobacillus salivarius PS2B (Active Comparator): Lactating women without mastitis (n=15)
  Interventions: Biological: Lactobacillus salivarius PS2

INTERVENTIONS:
Biological: Lactobacillus salivarius PS2 — 9.5 log10 (colony-forming units), freeze-dried powder, daily for 21 days
  Arms: Lactobacillus salivarius PS2
Biological: Lactobacillus salivarius PS2 — 9.5 log10 colony-forming units, oral route, freeze-dried powder, daily for 21 days
  Arms: Lactobacillus salivarius PS2B

SUMMARY:
In this study, the investigators will try to confirm if application of probiotic strains isolated from breast milk actually have a beneficial effect on women suffering lactational mastitis. This project has been design to offer an integrated vision of the effects of probiotherapy (Lactobacillus salivarius PS2) on the human host. Therefore, the investigators propose a multidisciplinary approach involving the application of microbiological, immunological, genomic, metagenomic, transcriptomic and metabolomic techniques. The hypothesis is that probiotherapy will cause different effects on the host, and the objective is the finding of markers that may support the beneficial effect of the strain in such condition.

ELIGIBILITY:
Inclusion Criteria:

* Normal term pregnancy
* Lactating women
* Healthy breastfed infant

Women with mastitis:

* Clinical symptoms of mastitis
* Painful breastfeeding
* Count of staphylococci, streptococci and/or corynebacteria in milk higher than 3,000 colony-forming units/mL
* Leukocyte count in milk higher 6 log10/mL

Women without mastitis:

* No clinical symptoms of mastitis
* No painful breastfeeding
* Count of staphylococci, streptococci and/or corynebacteria in milk lower than 500 colony-forming units/mL
* Leukocyte count in milk lower 5 log10/mL

Exclusion Criteria:

* Allergy to cow's milk protein
* Intolerance to lactose
* Antibiotic treatment
* Breast abscess
* Raynaud syndrome
* Any parallel disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Rodríguez, PhD, Study Director — Universidad Complutense de Madrid
Locations (1):
- Dpt. Nutricion, Bromatologia y Tecnologia de los Alimentos, Madrid, Madrid, Spain

REFERENCES:
- [Background] Arroyo R, Martin V, Maldonado A, Jimenez E, Fernandez L, Rodriguez JM. Treatment of infectious mastitis during lactation: antibiotics versus oral administration of Lactobacilli isolated from breast milk. Clin Infect Dis. 2010 Jun 15;50(12):1551-8. doi: 10.1086/652763. PMID 20455694
- [Background] Jimenez E, Fernandez L, Maldonado A, Martin R, Olivares M, Xaus J, Rodriguez JM. Oral administration of Lactobacillus strains isolated from breast milk as an alternative for the treatment of infectious mastitis during lactation. Appl Environ Microbiol. 2008 Aug;74(15):4650-5. doi: 10.1128/AEM.02599-07. Epub 2008 Jun 6. PMID 18539795
- [Result] Vazquez-Fresno R, Llorach R, Marinic J, Tulipani S, Garcia-Aloy M, Espinosa-Martos I, Jimenez E, Rodriguez JM, Andres-Lacueva C. Urinary metabolomic fingerprinting after consumption of a probiotic strain in women with mastitis. Pharmacol Res. 2014 Sep;87:160-5. doi: 10.1016/j.phrs.2014.05.010. Epub 2014 May 29. PMID 24880136

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactobacillus Salivarius PS2 | Lactobacillus Salivarius PS2B
Started | 25 | 15
Completed | 23 | 12
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: This study was designed to evaluate a high number of microbiological, biochemical or immunological parameters before and after the administration of a probiotic to women with mastitis and to elucidate which of them can be useful as biomarkers in future studies. The number of participants was considered suitable for such purpose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Salivarius PS2 | Lactobacillus Salivarius PS2B | Total
Number analyzed (Participants) | 25 | 15 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (7.7) | 29.0 (7.8) | 28.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 25 | 15 | 40
Total milk bacterial count (initial) [Mean (Standard Deviation); unit: log10 CFU/mL] | 4.08 (0.20) | 3.19 (0.59) | 3.63 (0.39)

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Clinically Definite Mastitis Confirmed by Microbiological Cultures and Somatic Cell Counts
Description: Total milk bacterial count at the end of the study (after probiotic administration for 21 days), measured as log10 of the number of colony-forming units per mL of milk
Time Frame: one week
Measure: Mean (95% Confidence Interval); unit: log10 CFU/mL
Arm/Group | Lactobacillus Salivarius PS2 | Lactobacillus Salivarius PS2B
Number analyzed (Participants) | 23 | 12
log10 CFU/mL | 3.09 [2.90 to 3.28] | 2.90 [2.12 to 3.70]

2. Secondary Outcome: Evidence of Changes in Gene Expression of Somatic Cells Obtained From Milk Samples
Time Frame: one year
Reporting Status: Not Posted

3. Secondary Outcome: Evidence of Changes in the Metabolic Profile of Urine
Time Frame: One year
Reporting Status: Not Posted

4. Secondary Outcome: Evidence of Changes in the Macronutrient and Electrolyte Profiles of Milk
Time Frame: One year
Reporting Status: Not Posted

5. Secondary Outcome: Evidence of Changes in the Immunological Profile of Milk
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Lactobacillus Salivarius PS2 | Lactobacillus Salivarius PS2B
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/15
Other Adverse Events (participants affected / at risk) | 0/25 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No